CLINICAL TRIAL: NCT03558347
Title: 5 Year Clinical Evaluation of CONELOG® Screw-Line Implants With 7 mm Length: a Prospective Randomized Double-blinded Clinical Study
Brief Title: CF41102 5-year Clinical Evaluation of Conelog® Implant With 7 mm Length
Acronym: UKAConelog
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: Camlog Oral Reconstruction Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKA 360569
Record Dates: First submitted 2018-05-04; First posted 2018-06-15 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Dental Implants; Partial Edentulism

STUDY DESIGN:
Intervention Model Description: This study consists of 20 patients (15 female, 5 male, mean age 59) who, after implant placement and second stage surgery, are randomly divided into two groups: group A was treated with two splinted crowns, group B with non-splinted single crowns. Four patients with bilateral free-end situation received both splinted and non-splinted restorations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short implants with splinted crowns (Experimental): Patients of that group received splinted crowns on the two adjacent implants Intervention: short implants with splinted crowns
  Interventions: Device: short implants with splinted crowns
- short implants with non-splinted crowns (Experimental): Patients of that group received single crowns on the two adjacent implants Intervention: short implants with non-splinted crowns
  Interventions: Device: short implants with non-splinted crowns

INTERVENTIONS:
Device: short implants with splinted crowns — 7 mm short implants (CONELOG® Implant System), individualized titanium abutments, splinted lithium disilicate crowns
  Other Names: CONELOG® Implant System
  Arms: short implants with splinted crowns
Device: short implants with non-splinted crowns — 7 mm short implants (CONELOG® Implant System), individualized titanium abutments, non-splinted lithium disilicate crowns
  Other Names: CONELOG® Implant System
  Arms: short implants with non-splinted crowns

SUMMARY:
The objective of this prospective, randomized, pilot study is to determine whether the Conelog® connection is suitable for splinted/non-splinted cemented crowns in the chewing centre (focus only on implant-abutment connection) and whether implants with the Conelog® connection and a length of 7mm are suitable for use in the molar region of the lower jaw.

DETAILED DESCRIPTION:
In order to avoid sinus augmentation in the upper jaw and a vertical augmentation in the lower jaw, various manufacturers offer short implants of 6-8mm length. The prevention of augmentative measures, especially in the mandible, is a fundamental component of the minimization of invasiveness while at the same time improving the functional capability. The benefit lies in the possibility to place implants without prior bone augmentation even in difficult anatomical conditions. This significantly reduces the invasiveness which on the one hand allows a higher number of patients to be treated with implants (especially morbid patients and anxiety patients) and on the other hand makes the treatment more predictable, with less risk, cost-efficient and considerably faster. Moreover, new scientific insights are gained in the area of short implants.

As with all implants, the risks associated with the study consist of intraoperative complications (e.g. damage of adjacent structures), failure of the implant (e.g. impairment of wound healing, fracture of the implant body), the abutment or abutment screw (e.g. loosening, fracture), or the crown on the abutment (veneer fracture, scaffold fracture).

The objective is to determine whether implants with the Conelog® connection and a length of 7mm are suitable for splinted/non-splinted monolithic lithium disilicate crowns cemented on individualized titanium abutments in the chewing centre of the mandible. The main indication for short implants is severe atrophy of the jaw, which creates a longer distance from the implant shoulder to the occlusal plane. An unfavourable crown-to-implant ratio means higher stress on the screws, the implant-abutment surface and possibly on the osseointegration of the implants. This raises the question whether splinted crowns have a positive effect on implant survival compared to non-splinted crowns.

The two 7mm Conelog ® implants are either used in the area of the second premolar and the first molar or the first and second molars of the mandible. The diameter of the implant depends on the width of the alveolar bone and ranges from 3.8 to 4.3 mm.

In case of a bilateral free-end situation, both quadrants are treated as part of the study, and both treatment variants are applied by using splinted crowns on one side and individual crowns on the other (split mouth design).

20 patients will be included in the study, which will be divided into two equally sized groups of 10 patients. All patients are recruited by the three clinical investigators at the Department of Prosthodontics and Biomaterials, Centre for Implantology, Medical Faculty, Rheinisch-Westfälische Technische Hochschule Aachen (RWTH) Aachen University Hospital. In order to achieve sufficient patient numbers, the population of Aachen will be informed via print media.

Each patient receives a single dose of antibiotics one hour prior to implant surgery. A mucoperiosteal flap was mobilized and the implants were placed as recommended by the manufacturer, using a surgical template as a guide. Healing abutments were screwed, and submerged healing is used for all implants. Second stage surgery is performed after 3 months. The prosthetic restoration is completed within 4 weeks after exposure.

Patients in group A will receive splinted monolithic lithium disilicate crowns cemented on individualized titanium abutments. Patients in group B will receive 2 non-splinted monolithic lithium disilicate-crowns cemented on individualized titanium abutments.

The cementation is done with Multilink Implant ® on the machined abutments, which have been cleaned for 5 minutes in an ultrasonic cleaner with 95% alcohol. The crowns are conditioned with hydrofluoric acid for 20 seconds and silanized with Monobond Plus® for 60 seconds. The day of insertion of the restoration is marked as baseline.

The examination performed at baseline and the follow up after 6 months includes occlusion, probing depth, plaque index and the condition of the ceramic surface of the crowns. Additionally, radiographs with customized positioning jigs are taken at baseline, after 1, 3, and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* female and male subjects older than 18 years
* absence of all molars and, optionally, the second premolar in at least on quadrant of the lower jaw
* the periodontal situation of the other teeth is healthy or periodontal treatment has already been successfully performed
* the antagonists are natural teeth or treated with fixed dentures
* good health according to the ASA Physical Status Classification System one or two (ASA 2010)
* good oral hygiene and an at most moderate tobacco consumption
* bone height above the N. alveolaris inferior of at least 11mm and the precondition of a one-stage implantation and augmentation
* signed consent

Exclusion Criteria:

* Indication for large augmentations of the jaw bone
* Bone abundance with minimal risk of injury to neighbouring structures when using two 11 mm or longer implants
* Psychological disorder
* substance abuse
* removable dentures (with or without implants)
* pregnancy
* patients under age or unable to reason
* persons who are placed in an institution on a judicial or administrative order

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2021-09-27 (Estimated)

PRIMARY OUTCOMES:
marginal bone loss | 5 years
  measurement of marginal bone loss on standardized radiographs [mm]

SECONDARY OUTCOMES:
probing depth | 5 years
  measurement of probing depth [mm]
gingival status | 5 years
  assessment of gingival index
oral hygiene | 5 years
  assessment of plaque index
survival rate of prosthetic restoration | 5 years
  screw loosening, screw fracture, implant fracture, chippings

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Wolfart, Prof. Dr., Study Director — University Hospital, Aachen
Locations (1):
- Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tawil G, Aboujaoude N, Younan R. Influence of prosthetic parameters on the survival and complication rates of short implants. Int J Oral Maxillofac Implants. 2006 Mar-Apr;21(2):275-82. PMID 16634499
- [Background] Misch CE. Short dental implants: a literature review and rationale for use. Dent Today. 2005 Aug;24(8):64-6, 68. PMID 16161821
- [Background] Vehemente VA, Chuang SK, Daher S, Muftu A, Dodson TB. Risk factors affecting dental implant survival. J Oral Implantol. 2002;28(2):74-81. doi: 10.1563/1548-1336(2002)0282.3.CO;2. PMID 12498449
- [Background] Gentile MA, Chuang SK, Dodson TB. Survival estimates and risk factors for failure with 6 x 5.7-mm implants. Int J Oral Maxillofac Implants. 2005 Nov-Dec;20(6):930-7. PMID 16392351
- [Background] Urdaneta RA, Rodriguez S, McNeil DC, Weed M, Chuang SK. The effect of increased crown-to-implant ratio on single-tooth locking-taper implants. Int J Oral Maxillofac Implants. 2010 Jul-Aug;25(4):729-43. PMID 20657868
- [Background] Li R, Sun W, Shi B. [Retrospective analysis of placing short dental implants in the posterior areas]. Zhonghua Kou Qiang Yi Xue Za Zhi. 2010 Dec;45(12):708-11. Chinese. PMID 21211233
- [Background] Yi YS, Emanuel KM, Chuang SK. Short (5.0 x 5.0 mm) implant placements and restoration with integrated abutment crowns. Implant Dent. 2011 Apr;20(2):125-30. doi: 10.1097/ID.0b013e31820fb67e. PMID 21448021
- [Background] Etoz OA, Ulu M, Kesim B. Treatment of patient with Papillon-Lefevre syndrome with short dental implants: a case report. Implant Dent. 2010 Oct;19(5):394-9. doi: 10.1097/ID.0b013e3181ed0798. PMID 20881810
- [Background] Ogawa T, Dhaliwal S, Naert I, Mine A, Kronstrom M, Sasaki K, Duyck J. Effect of tilted and short distal implants on axial forces and bending moments in implants supporting fixed dental prostheses: an in vitro study. Int J Prosthodont. 2010 Nov-Dec;23(6):566-73. PMID 21209995
- [Background] Wu H, Li JH, DI P, Qiu LX, Lin Y, Luo J. [A long-term retrospective clinical study of short dental implant restoration]. Zhonghua Kou Qiang Yi Xue Za Zhi. 2010 Dec;45(12):712-6. Chinese. PMID 21211234
- [Background] De Santis D, Cucchi A, Longhi C, Vincenzo B. Short threaded implants with an oxidized surface to restore posterior teeth: 1- to 3-year results of a prospective study. Int J Oral Maxillofac Implants. 2011 Mar-Apr;26(2):393-403. PMID 21483893
- [Background] Neldam CA, Pinholt EM. State of the art of short dental implants: a systematic review of the literature. Clin Implant Dent Relat Res. 2012 Aug;14(4):622-32. doi: 10.1111/j.1708-8208.2010.00303.x. Epub 2010 Oct 26. PMID 20977606
- [Background] Raviv E, Turcotte A, Harel-Raviv M. Short dental implants in reduced alveolar bone height. Quintessence Int. 2010 Jul-Aug;41(7):575-9. PMID 20614044
- [Background] Hasan I, Heinemann F, Aitlahrach M, Bourauel C. Biomechanical finite element analysis of small diameter and short dental implant. Biomed Tech (Berl). 2010 Dec;55(6):341-50. doi: 10.1515/BMT.2010.049. Epub 2010 Oct 28. PMID 21028950
- [Derived] Al-Sawaf O, Tuna T, Rittich A, Kern T, Wolfart S. Randomized clinical trial evaluating the effect of splinting crowns on short implants in the mandible 3 years after loading. Clin Oral Implants Res. 2020 Nov;31(11):1061-1071. doi: 10.1111/clr.13652. Epub 2020 Sep 12. PMID 33463774